CLINICAL TRIAL: NCT03589859
Title: Computerized Game-based Vestibular Rehabilitation: Assessment of Feasibility and Motor Learning
Brief Title: Computerized Vestibular Rehabilitation
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: C2892-P
Record Dates: First submitted 2018-07-06; First posted 2018-07-18 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-10

CONDITIONS: Vestibular Diseases
Keywords: neurologic rehabilitation; computer games
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — No biological specimens will be retained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Normal Volunteers: Testing motor learning
  Interventions: Diagnostic Test: VOR Test; Other: Computer Game
- Vestibular hypofunction: Testing feasibility of rehabilitation game
  Interventions: Diagnostic Test: VOR Test; Other: Computer Game; Other: Nausea Scale

INTERVENTIONS:
Diagnostic Test: VOR Test — Video-oculography is used to record the vestibulo-ocular reflex during active and passive turns of the head.
Other: Computer Game — Participants play a custom computer game that is designed to produce motor learning in the vestibulo-ocular reflex
Other: Nausea Scale — Participants asked to rate their subjective nausea on a numeric scale after playing units of the computer game
  Groups: Vestibular hypofunction

SUMMARY:
Disorders of vestibular function and balance are an important component of many conditions that commonly affect veterans, such as inner ear diseases, diabetes, and traumatic brain injury. Veterans with vestibular impairment have reduced quality of life, limitations on work and physical activities, and an increased risk of falls. The goal of this research is to develop a more engaging and effective interactive tool for vestibular rehabilitation to improve the lives of affected veterans. The first steps in this process will be to test the ability of the application to facilitate vestibular learning and to test its feasibility in vestibular patients. The hypothesis is that computer-game-based adaptation will induce robust VOR motor learning and will provide an engaging platform for vestibular rehabilitation. Ultimately, our application has the potential to provide more flexible vestibular exercises that will allow therapy to be customized for each patient. It will also have the ability to track a patient's progress over time and to advance exercises as function improves.

ELIGIBILITY:
Inclusion Criteria:

* GROUP 1: Healthy volunteers: Static visual acuity of at least 20/30 at testing distance
* GROUP 2: Vestibular patients: Unilateral or bilateral vestibular hypofunction, No central vestibular disorder, Static Visual Acuity of at least 20/30 at testing distance

Exclusion Criteria:

* GROUP 1: Peripheral or central vestibular disorder
* GROUP 2: Central vestibular disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal volunteers and patients with vestibular hypofunction
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark F. Walker, MD, Principal Investigator — Louis Stokes VA Medical Center, Cleveland, OH
Locations (1):
- Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
A limited set of de-identified data supporting published results will be made available on request, pursuant to a Data Use Agreement.
Time Frame: Pursuant to Data Use Agreement
Access Criteria: Pursuant to Data Use Agreement

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Volunteers: Healthy individuals with intact vestibular function
  VOR Test: Video-oculography is used to record the vestibulo-ocular reflex during active and passive turns of the head.
  Computer Game: Participants play a custom computer game that is designed to produce motor learning in the vestibulo-ocular reflex
- Vestibular Hypofunction: Veterans with peripheral vestibular hypofunction
  VOR Test: Video-oculography is used to record the vestibulo-ocular reflex during active and passive turns of the head.
  Computer Game: Participants play a custom computer game that is designed to produce motor learning in the vestibulo-ocular reflex
Period: Overall Study
Arm/Group | Normal Volunteers | Vestibular Hypofunction
Started | 18 | 6
Completed | 18 | 0
Not Completed | 0 | 6
Not completed — Withdrawal by Subject | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Volunteers | Vestibular Hypofunction | Total
Number analyzed (Participants) | 18 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (13) | 61 (15) | 42 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 0 | 9
  Male | 9 | 6 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 16 | 6 | 22
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 14 | 5 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 6 | 24
Dizziness Handicap Inventory [Mean (Standard Deviation); unit: units on a scale] — The Dizziness Handicap Inventory is a 25-item questionnaire that has a score range of 0-100. Higher scores mean worse dizziness. Population: Assessed only in participants with vestibular dysfunction
  units on a scale
    number analyzed (Participants) | 0 | 6 | 6
    (all) |  | 31.6 (16.7) | 31.6 (16.7)
Activities-specific Balance Confidence scale [Mean (Standard Deviation); unit: units on a scale] — The Activities-Balance Confidence Scale is a 16-item questionnaire that assesses an individual's confidence in doing various activities that require balance. Each is given a percentage from 0% to 100% confidence in performing that activity. The number reported is the mean of these individual percentages. Higher numbers mean more confidence (better). Population: Assessed only in participants with vestibular dysfunction
  units on a scale
    number analyzed (Participants) | 0 | 6 | 6
    (all) |  | 79.5 (14.0) | 79.5 (14.0)

OUTCOME MEASURES:

1. Primary Outcome: Vestibulo-ocular Reflex Gain Ratio
Description: The vestibulo-ocular reflex gain is the relationship between a rotation of the head and the evoked eye movement. The outcome measure is the ratio of the VOR gain after training to that before training. VOR gain is determined by a scaled fit of eye speed to evoking head speed (normal gain is 1). Note that this experiment was not a treatment of impairment but a test of the ability of the vestibular game to elicit motor learning (away from normal) in individuals with intact motor learning. In that context, an increase in the gain to a value greater than unity (faster eye movement relative to the head movement) is "better" with respect to the training goal, but it is not "better" with respect to real-world visual function, for which a gain of one is the goal. There is no threshold value for this type of motor learning experiment. Instead, the question is whether the gain is increased after training, and if so, by what percentage relative to the training goal.
Time Frame: VOR measurements to determine gain were performed immediately before and after each approximately 30 minute training session. Pre- and post-training gains were then combined in the VOR gain ratio to determine the training effect.
Population: This measure applied only to Group 1: healthy individuals with intact vestibular function
Measure: Mean (95% Confidence Interval); unit: unitless gain ratio
Groups:
- Vestibular Hypofunction: Veterans with vestibular hypofunction
Arm/Group | Normal Volunteers | Vestibular Hypofunction
Number analyzed (Participants) | 18 | 0
unitless gain ratio | 1.15 [1.10 to 1.20] |
Statistical Analysis 1: Comparison: Normal Volunteers; A linear mixed effects model was used to compare pre- and post-training VOR gains; Test type: Other — This was a physiology study, not a treatment trial. The test was for a change in VOR gain; p < 0.001, Mixed Models Analysis

2. Other Pre Specified Outcome: Nausea Scale
Description: Participants with vestibular hypofunction rated their nausea after each game block on a scale of 1 to 10. For each visit, there were up to 3 game-blocks, each of 10-minutes duration. The number of blocks was determined by the participant. A higher score is a worse outcome (more nausea). The average nausea scale rating was determined for each participant. The final result is the median of these averaged scores.
Time Frame: Immediately after each 10-minute game block, median value calculated for each participant
Population: This measure applied only to Group 2: participants with vestibular dysfunction. Of the 6 enrolled participants in this group, one chose not to complete the game playing after consenting, and a second was found to have recovery of his vestibular function before game playing. The reported data are from the remaining four participants.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Normal Volunteers | Vestibular Hypofunction
Number analyzed (Participants) | 0 | 4
score on a scale |  | 1.2 [0 to 4.5]

ADVERSE EVENTS:
Time Frame: For the full duration of the study (4 years).
Description: The procedure was to report adverse events to the local IRB.
Arm/Group | Normal Volunteers | Vestibular Hypofunction
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/6
Other Adverse Events (participants affected / at risk) | 0/18 | 0/6

LIMITATIONS AND CAVEATS:
No conclusions can be made regarding the therapeutic efficacy of the computer game for treatment of vestibular hypofunction, because the study was not designed to test that. Instead, its objectives were, first, to test the game's ability to induce motor learning, to establish a physiological basis for therapeutic use, and, second, to test feasibility and playability by individuals with vestibular disorders.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-04): https://cdn.clinicaltrials.gov/large-docs/59/NCT03589859/Prot_SAP_000.pdf